CLINICAL TRIAL: NCT02736175
Title: A Prospective, Multicenter, Randomized, Parallel-Arm, Double-Masked, Vehicle Controlled Phase 3C Study Evaluating the Safety and Efficacy of OTX-DP for the Treatment of Ocular Inflammation and Pain After Cataract Surgery
Brief Title: OTX-15:003: A Phase 3 Study Evaluating the Safety and Efficacy of OTX-DP for the Treatment of Ocular Inflammation and Pain After Cataract Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ocular Therapeutix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OTX-15-003
Record Dates: First submitted 2016-02-10; First posted 2016-04-13 (Estimated); Results first posted 2017-10-11 (Actual); Last update posted 2017-11-13 (Actual); Status verified 2017-10

CONDITIONS: Post-Surgical Ocular Pain; Post-Surgical Ocular Inflammation
MeSH Terms: interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- OTX-DP (Experimental): OTX-DP (dexamethasone insert) 0.4 mg for intracanalicular use
  Interventions: Drug: Dexamethasone
- PV (Placebo Comparator): PV (placebo drug delivery vehicle)
  Interventions: Other: Placebo Vehicle

INTERVENTIONS:
Drug: Dexamethasone
  Arms: OTX-DP
Other: Placebo Vehicle
  Arms: PV

SUMMARY:
The objective of the study was to evaluate the safety and efficacy of OTX-DP (dexamethasone insert) 0.4 mg for intracanalicular use when placed in the canaliculus of the eyelid for the treatment of post-surgical inflammation and pain in subjects who had undergone cataract extraction with intraocular lens implantation

ELIGIBILITY:
Inclusion Criteria:

* Has a cataract and is expected to undergo clear corneal cataract surgery with phacoemulsification and implantation of posterior chamber lens
* Has a potential post-operative pinhole corrected Snellen VA of at least 20/200 or better in both eyes

Exclusion Criteria:

* Any intraocular inflammation in the study eye present during the screening slit lamp examination
* Score greater than "0" on the Ocular Pain Assessment in the study eye at Screening
* Any intraocular inflammation in the study eye present during the screening slit lamp examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 438 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-07 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Vehicle: PV (placebo drug delivery vehicle)
Period: Overall Study
Arm/Group | OTX-DP | Placebo Vehicle
Started | 216 | 222
Completed | 214 | 221
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Population: All randomized subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | OTX-DP | Placebo Vehicle | Total
Number analyzed (Participants) | 216 | 222 | 438
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (9.09) | 68.6 (8.37) | 68.0 (8.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120 | 130 | 250
  Male | 96 | 92 | 188
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 37 | 37 | 74
  Not Hispanic or Latino | 179 | 185 | 364
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 8 | 1 | 9
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 28 | 25 | 53
  White | 174 | 189 | 363
  More than one race | NA — Not collected in this manner | NA — Not collected in this manner | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported | 3 | 4 | 7
Iris Color [Count of Participants; unit: Participants]
  Brown | 106 | 101 | 207
  Blue | 61 | 64 | 125
  Hazel | 32 | 37 | 69
  Green | 15 | 18 | 33
  Gray | 2 | 0 | 2
  Black | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Absence of Anterior Chamber Inflammation
Description: Absence of cells (i.e., score of '0') in the anterior chamber of the study eye at Day 14
Time Frame: Day 14
Population: ITT LOCF (last observation carried forward)
Measure: Number; unit: percentage of total participants
Arm/Group | OTX-DP | Placebo Vehicle
Number analyzed (Participants) | 216 | 222
percentage of total participants | 52.3 | 31.1

2. Primary Outcome: Absence of Ocular Pain
Description: Absence of pain (i.e., score of '0') in the study eye at Day 8
Time Frame: Day 8
Population: ITT LOCF (last observation carried forward)
Measure: Number; unit: percentage of total participants
Arm/Group | OTX-DP | Placebo Vehicle
Number analyzed (Participants) | 216 | 222
percentage of total participants | 79.6 | 61.3

ADVERSE EVENTS:
Arm/Group | OTX-DP | Placebo Vehicle
All-Cause Mortality (participants affected / at risk) | 0/216 | 0/221
Serious Adverse Events (participants affected / at risk) | 3/216 | 2/221
Other Adverse Events (participants affected / at risk) | 63/216 | 86/221
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OTX-DP (N=216) | Placebo Vehicle (N=221)
Retinal detachment (Eye disorders) | 1 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OTX-DP (N=216) | Placebo Vehicle (N=221)
Adverse Events (General disorders) | 63 (91) | 86 (109)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No